CLINICAL TRIAL: NCT00178737
Title: Does the Message Matter? Enhancing Adherence in Healthcare Through Persuasive Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSC-SHIS-05-0240
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Appointment Reminders

INTERVENTIONS:
Behavioral: Electronic reminder message

SUMMARY:
In this research we propose to develop a comprehensive model to explain how users process persuasive messages. We then propose to experimentally test varying the persuasiveness of message content in various domains, and assess their impact on adherence by both physicians and patients. Finally based on our conceptual model and results from the experimental data we propose to develop preliminary guidelines to assist developers in designing effective messages.

ELIGIBILITY:
Inclusion Criteria:

Study 1

1. Subjects who have an appointment scheduled at HCHD Baytown Health Center

Study 2

1. Subjects who are neonatology physicians (not in training).
2. Subjects must be able to give signed informed consent.

Study 3

1. Any subjects (students or employee) at the University of Texas Health Science Center at Houston.
2. Subjects must be able to give signed informed consent.

Exclusion Criteria:

* No specific individual who meets the inclusion criteria will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad F Walji, M.S., Principal Investigator — The University of Texas Health Science Center, Houston